CLINICAL TRIAL: NCT04727398
Title: The Incidence of Complete Posterior Vitreous Degeneration After Phacoemulsification
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Suthasinee Sinawat, Associate Professor, Khon Kaen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HE631092
Record Dates: First submitted 2021-01-24; First posted 2021-01-27 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Posterior Vitreous Detachment
Keywords: posterior vitreous detachment; phacoemulsification
MeSH Terms: conditions — Vitreous Detachment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cataract patients who was scheduled for phacoemulsification (Other): Wide-field optical coherence tomography was performed before the surgery, and then was done at 1, 3, 6 and 12 months following the phacoemulsification.
  Interventions: Device: Wide-field optical coherence tomography (Optovue®)

INTERVENTIONS:
Device: Wide-field optical coherence tomography (Optovue®) — Merged 4 images for wide-filed OCT-based PVD classification, 2 vertical line images and 2 horizontal line images

SUMMARY:
Intraocular surgery could induce vitreous degeneration and then abnormal posterior vitreous detachment (PVD) could occur including vitreoschisis and partial-thickness PVD. Vitreomacular interface (VMI) abnormalities such as epimacular membrane were observed following many intraocular surgeries. The incidence of peripheral break and epimacular membrane (EMM) after pneumatic retinopexy were 11.7% and 4-11%, respectively. Although multiple intravitreal anti-vascular endothelial growth factor (anti-VEGF) injections induced PVD of 5.6%, but peripheral break was reported as only 0.67%. The incidence of rhegmatogenous retinal detachment (RRD) after phacoemulsification is gradually increased with time. The accumulative risk of RRD was increased from 0.27% at 1 year to 1.27% at 20 years after phacoemulsification.

DETAILED DESCRIPTION:
The most common intraocular surgery is cataract surgery. From the literature review, many methods were used to detect the PVD after phacoemulsification. The former studies used indirect ophthalmoscopy and ocular ultrasound for diagnosis of PVD. The later studies used the optical coherence tomography (OCT) for PVD detection. The OCT device had higher effectiveness in evaluation of the posterior segment, and then it can detect post-phacoemulsification PVD more and early than previous studies. Ivastinovic et al demonstrated 59.2% of patients had PVD at 1 month after phacoemulsification, and increased up to 71.4% at 3 months.

Tsukahara et al introduced wide-field OCT-based PVD classification. The advance OCT device will be useful in detection of abnormal PVD and it's sequelae. If the risk factors of post-phacoemulsification PVD were explored, the prevention of abnormal PVD and VMI disorders could be done.

ELIGIBILITY:
Inclusion Criteria:

* Cataract patients who was scheduled for phacoemulsification
* Age >50 years
* No complete PVD was detected by OCT
* Can be taken the wide-field OCT images
* Written informed consent

Exclusion Criteria:

* Secondary cataract)
* History of ocular trauma or head trauma
* Systemic diseases that can cause the intraocular problems such as connective tissue disease
* History of other ocular diseases such as glaucoma, uveitis and vitreoretinal disorders
* History of intraocular laser treatment
* History of intraocular surgery such as intravitreal drug injection

Withdrawal Criteria:

* Intraoperative complications such as posterior capsular rupture and zonule dialysis
* Postoperative complications such as vitreous hemorrhage and postoperative endophthalmitis
* Undergo the intraocular surgery during the follow-up period
* Receiving the intraocular laser treatment during the follow-up period such as laser capsulotomy and panretinal photocoagulation
* Having the ocular trauma or head trauma during the follow-up period

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2021-09-03 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of PVD after phacoemulsification | 12 months
  incidence of complete PVD

SECONDARY OUTCOMES:
The incidence of VMI disorders | 12 months
  e.g. Epimacular membrane, Vitreomacular traction, Peripheral retinal break

CONTACTS AND LOCATIONS:
Overall Officials: Suthasinee Sinawat, MD, Principal Investigator — KKU Eye Center, Department of Ophthalmology, Faculty of Medicine, Khon Kaen University
Locations (1):
- Khon Kaen University, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No